CLINICAL TRIAL: NCT02675816
Title: Inspire® Upper Airway Stimulation System: Randomized Control Trial / European Post-Market Study
Brief Title: Inspire® Upper Airway Stimulation System
Acronym: RCT
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Study halted due to low recruitment. Reimbursement changes require a larger study with additional centers and therefore, a new study planned as replacement.
Sponsor: Inspire Medical Systems, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2015-001
Record Dates: First submitted 2016-01-28; First posted 2016-02-05 (Estimated); Last update posted 2016-08-11 (Estimated); Status verified 2016-08

CONDITIONS: Obstructive Sleep Apnea
Keywords: Obstructive Sleep Apnea; OSA; neurostimulation; hypoglossal nerve; tongue; upper airway stimulation; surgery
MeSH Terms: conditions — Sleep Apnea, Obstructive | interventions — Drug Delivery Systems

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Inspire® (UAS) System (Other): This is a single-arm study; all participants will be implanted with the Inspire® Upper Airway Stimulation (UAS) System.
  Interventions: Device: Inspire® Upper Airway Stimulation (UAS) System

INTERVENTIONS:
Device: Inspire® Upper Airway Stimulation (UAS) System — This is a single-arm study; all participants will be implanted with the Inspire® Upper Airway Stimulation (UAS) System. This is a permanent, implantable therapy device, which consists of three implantable components: an implantable pulse generator (IPG), a stimulation lead, and a sensing lead. In addition, the patient receives a handheld remote to activate the therapy
  Other Names: Inspire® Therapy

SUMMARY:
The purpose of this post-market study is to assess safety and effectiveness of Inspire Upper Airway System (UAS) in a commercial setting. This study will provide additional clinical evidence of Inspire UAS for treatment of moderate to severe obstructive sleep apnea (OSA) using a randomized controlled trial design.

DETAILED DESCRIPTION:
This study is a prospective, multi-center, randomized controlled study with a delayed start arm, conducted under a common implant protocol.

Up to 40 study subjects will be implanted at up to six centers in Europe. Subjects will be evaluated at baseline, implant, post-op (randomized) and 1-, 2-, 3,- 4- and 6-months post-implant.

Baseline data will include collection of demographics and medical history, completion of a physical exam, Functional Tongue Exam (FTE), and subject quality of life (QoL) questionnaires (Functional Outcomes of Sleep Questionnaire (FOSQ) and Epworth Sleepiness Scale (ESS)). Adverse event data will be collected from the time of baseline testing through the 6-month study follow-up.

Implant eligibility assessments will include home sleep testing (HST), a surgical consultation and a drug induced sedated endoscopy (DISE) to determine if the subject is a qualified candidate for implant.

Subjects meeting all baseline and pre-screening requirements will be implanted with the Inspire system. Intra- and post- operative procedure data will be collected. Subjects will be seen for a post-operative check one week after implant. During this visit, subjects will be randomized 1:1 to the ACTIVE group or the DELAY group. However, the Inspire system will not be activated (turned "on") during the first month post-implant to allow for post-surgical healing.

Only subjects randomized to the ACTIVE group will return for the 1-month follow-up visit at which time the device will be activated (turned "on"). The subjects will be provided with a patient remote and instructed on its use. These ACTIVE arm subjects will be instructed to use their Inspire system on a nightly basis and return for a 2-month visit for an in-laboratory sleep study to complete device titration.

All subjects (ACTIVE and DELAY) return for the 3-month visit to complete a HST (DELAY subjects' therapy will remain off during the HST). In addition, QoL and patient satisfaction surveys, Functional Tongue Exam (FTE), and general health assessments, including adverse event review, will be collected. Subjects in the DELAY arm will have their therapy activated at the end of the 3 month visit, and return for a 4-month visit for an in-laboratory sleep study to complete device titration. All subjects will return for a 6-month and final visit where a two-night HST will be completed. In addition, QoL and patient satisfaction surveys, physical exam and FTE data will be collected; a device check will be completed as well as adverse event review. Therapy usage and device adjustment data, as well as a subject satisfaction with therapy survey, will be collected for additional analysis. Safety data will be collected throughout the study.

ELIGIBILITY:
Inclusion Criteria:

1. Meet the requirements per current CE Mark labeling
2. Willing and capable to have stimulation hardware permanently implanted, and to use the patient remote to activate the stimulation
3. Willing and capable to return for all follow-up visits and conduct sleep studies at home, including the evaluation procedures and filling out questionnaires
4. Willing and capable of providing informed consent

Exclusion Criteria:

1. Do not meet any contraindications per current CE Mark labeling
2. Body Mass Index (BMI) of > 35
3. Central + mixed apneas > 25% of the total apnea-hypopnea index (AHI)
4. Any chronic medical illness or condition that contraindicates a surgical procedure under general anesthesia, as judged by the clinical study Investigator
5. Has a terminal illness with life expectancy < 12 months
6. Active psychiatric disease (psychotic illness, major depression, or acute anxiety attacks) which prevents subject compliance with the requirements of the investigational study testing
7. Any other reason the investigator deems subject is unfit for participation in the study

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2015-08; Primary Completion 2016-07 (Actual); Study Completion 2016-07 (Actual)

PRIMARY OUTCOMES:
Change from Baseline OSA at 3 Months | 3 months post-implant
  The percent of apnea hypopnea index (AHI) reduction will be used as a primary endpoint to quantify the effects of the Inspire therapy on OSA between the 'Active' therapy (ACTIVE) and 'Delayed Start' therapy (DELAY). The percent of AHI reduction is the percent change between baseline AHI at the pre-implant sleep study and AHI at the 3-month post-implant sleep study.

SECONDARY OUTCOMES:
Number of Reported SAEs / Procedure & Device Related AEs | 6 months post-implant
  Safety of the therapy will be assessed via the description of all reported SAEs and all procedure- or device-related AEs. Adverse events will be summarized by seriousness, severity, relatedness to the device and/or procedure and temporal relationship to the procedure. No formal statistical hypotheses will be tested. Only device- or procedure-related AEs will be collected in this post-market study.
Change from Baseline OSA at 6 Months | 6 months post-implant
  AHI at the 6-month follow-up will be compared to the AHI at baseline in both the ACTIVE and DELAY groups.
Change from Baseline Breathing Indices at 6 Months | 6 months post-implant
  Sleep disordered breathing indices at the 6-month follow-up will be compared to the breathing indices at baseline.
Change from Baseline Quality of Life Questionnaires (QoL) | 6 months post-implant
  Quality of Life (QoL) questionnaires at the 6-month visit will be compared to the QoL questionnaires at baseline.

CONTACTS AND LOCATIONS:
Overall Officials: Clemens Heiser, Dr. med., Principal Investigator — Klinikum rechts der Isar der Technischen Universität München; Joachim T Maurer, OA Dr. med., Principal Investigator — Universitäts-HNO-Klinik Mannheim; Armin Steffen, PD Dr. med., Principal Investigator — Klinik für HNO-Heilkunde/HNO-Schlaflabor; Olivier Vanderveken, Prof. dr., Principal Investigator — University Hospital, Antwerp
Locations (4):
- Universitair Ziekenhuis Antwerpen, Antwerp, Belgium
- Germany (3):
  - Klinik für HNO-Heilkunde/HNO-Schlaflabor, Lübeck
  - Universitäts-HNO-Klinik Mannheim, Mannheim
  - Klinikum rechts der Isar der Technischen Universität München, München

IPD SHARING:
Plan to Share IPD: Yes